CLINICAL TRIAL: NCT01030744
Title: Evaluation of the Gestational Diabetes Self-Management Education Program and Quality Improvement Plan
Acronym: GDM Elasy
Status: Withdrawn | Type: Observational
Why Stopped: This is quality improvement review and should not have been registered. No participants were enrolled
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: GDM Elasy
Record Dates: First submitted 2009-11-30; First posted 2009-12-11 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Self-Monitoring of Blood Glucose
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gestational Diabetes: Women with gestational diabetes who are referred to and followed in the Vanderbilt Eskind Diabetes Clinic and are participants in the gestational diabetes educational program.

SUMMARY:
The broad, long-term objectives are to generate and test hypotheses leading to theories that guide improved care of patients with gestational diabetes. The purpose of this chart review study is to evaluate the Vanderbilt Gestational Diabetes Self-Management Education Program and Quality Improvement Plan in optimizing metabolic control and improving health outcomes during pregnancy with gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Women with gestational diabetes who are referred to and followed in the Vanderbilt Eskind Diabetes Clinic and are participants in the gestational diabetes educational program.

Exclusion Criteria:

* Refusal of consent.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with gestational diabetes who are referred to and followed in the Vanderbilt Eskind Diabetes Clinic and are participants in the gestational diabetes educational program.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Self-Monitoring of Blood Glucose | chart review quarterly during course of study

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University : Vanderbilt Diabetes Center (VDC), Nashville, Tennessee, United States